CLINICAL TRIAL: NCT02287077
Title: A Randomized Controlled Trial of Umbilical Cord Milking for Neonates With Hypoxic Ischemic Encephalopathy
Brief Title: Umbilical Cord Milking for Neonates With Hypoxic Ischemic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Lata Mangeshkar Hospital, NKP Salve Institute of Medical Sciences, Nagpur, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14D.522
Record Dates: First submitted 2014-10-31; First posted 2014-11-10 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Hypoxic Ischemic Encephalopathy; Umbilical Cord Milking
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate cord clamping (No Intervention): At birth, neonate will be held at the level of placenta and umbilical cord will be clamped immediately (standard of care for depressed neonates).
- Umbilical cord milking (Experimental): At birth, neonate will be held below the level of placenta and umbilical cord will be milked 3 times before clamping the cord.
  Interventions: Procedure: Umbilical Cord Milking

INTERVENTIONS:
Procedure: Umbilical Cord Milking — At birth, neonate will be held below the level of placenta and umbilical cord will be milked 3 times before clamping the cord.
  Other Names: Umbilical cord stripping
  Arms: Umbilical cord milking

SUMMARY:
The objective of this pilot study is to investigate the feasibility of performing umbilical cord milking in neonates who are depressed at birth.

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy (HIE) is a brain injury in neonates due to inadequate blood flow and oxygen delivery to the neonatal brain. Umbilical cord milking can potentially improve brain injury in neonates with HIE. The objective of this study is to investigate the feasibility of performing umbilical cord milking in neonates who are depressed at birth. The investigators hypothesized that umbilical cord milking is feasible and safe in neonates who are depressed at birth. The investigators also hypothesized that umbilical cord milking will increase stem cells in neonatal blood circulation and improve short term outcomes in neonates with moderate and severe HIE.

ELIGIBILITY:
Inclusion Criteria:

* Term and near term neonates (35 weeks and more)
* Depressed at birth

Exclusion Criteria:

* Congenital malformation of central nervous system
* Chromosomal abnormalities
* Major congenital malformations

Max Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2014-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The number of depressed neonates in whom umbilical cord milking was performed. | Participants will be followed for the duration of hospital stay, an expected average of 5 days
  The number of neonates who are depressed at birth will be determined and the percentage of depressed neonates in whom UCM performed will be calculated. The investigators expect that more than 80% of neonates who qualify will receive UCM. The investigators will aslo compare resuscitation efforts (use of positive pressure ventilation, intubation, chest compression, medication and fluid boluses) and short term outcomes of resuscitation (5 minutes apgar, severity of HIE, blood gas at 1 hour) in neonates with and without UCM.

SECONDARY OUTCOMES:
The effect of umbilical cord milking on stem and progenitor cells in peripheral blood of neonates. | 24 hours
  Evaluate stem and progenitor cell count in peripheral blood of neonates with UCM and compare them with the control group (no UCM).
The effect of umbilical cord milking on monocytes and lymphocytes in peripheral blood of neonates. | 24 hours
  Evaluate absolute monocyte and lymphocyte count in peripheral blood of neonates with UCM and compare them with the control group (no UCM).
The effect of umbilical cord milking on neurotrophic factors in peripheral blood of neonates. | 24 hours
  Compare levels of neurotrophic factors in peripheral blood of neonates with and without UCM.
Survival and short term outcomes in neonates with moderate and severe HIE | Participants will be followed for the duration of hospital stay, an expected average of 5 days
  In infants with moderate or severe HIE, compare survival, neurological examination at discharge, and neuro-imaging studies in infants with and without UCM.

CONTACTS AND LOCATIONS:
Locations (1):
- Lata Mangeshkar Hospital and NKP Salve Institute of Medical Sciences, Nagpur, MS, India